CLINICAL TRIAL: NCT07149961
Title: Supplementation of Piperine and Curcumin (Curcuma Xanthorrhiza) Extract in ST Elevation Myocardial Infarction - SPICE STEMI Trial
Brief Title: Curcumin-Piperine Supplementation in STEMI - SPICE STEMI Trial
Acronym: SPICE STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Collaborators: Dr. Kariadi Hospital Semarang, indonesia (Unknown)
Responsible Party: Principal Investigator, Fahri Husaini Alkaf, dr. Fahri Husaini Alkaf, M.H., Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 984/UN7.F4/PP/II/2025; 984/UN7.F4/PP/II/2025 (Other Grant/Funding Number: Universitas Diponegoro)
Record Dates: First submitted 2025-08-16; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: ST Elevation Myocardial Infarction (STEMI); Malondialdehyde; Hs-CRP; Curcumin; Curcuma Xanthorrhiza; High-sensitivity C-reactive Protein
Keywords: Curcumin; Piperine; Turmeric (Curcuma Xanthorrhiza); Piper nigrum; ST Elevation Myocardial Infarction; Primary Percutaneous Coronary Intervention (PPCI); Oxidative Stress; Inflammation; High-sensitivity C-Reactive Protein; Malondialdehyde; Antioxidants; Anti-Inflammatory Agents
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Inflammation | interventions — Curcumin; piperine; turmeric extract

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to receive either curcumin-piperine supplementation or matching placebo, administered daily for 28 days following primary percutaneous coronary intervention for STEMI. Both groups are followed in parallel for the same duration, with biomarker measurements taken at baseline, 48-72 hours post-procedure, and at day 28.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcomes assessors are unaware of group allocation. Placebo capsules are identical in appearance, size, and packaging to the curcumin-piperine capsules to maintain blinding. Randomization codes are kept by an independent pharmacist until data analysis is complete.
  An independent pharmacist and data analyst are also masked to group allocation until database lock. Laboratory personnel performing biomarker analyses (hsCRP and MDA) are blinded to treatment assignment. Randomization codes are securely stored and only accessible to an independent statistician not involved in patient care or outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants receive a matching placebo capsule identical in appearance, size, and packaging to the curcumin-piperine capsule, administered daily for 28 consecutive days following PPCI for STEMI. A loading dose of 2 placebo capsules is administered orally prior to PPCI, followed by maintenance of 1 capsule twice daily until day 28.
  Interventions: Other: Placebo capsules
- Curcumin-Piperine Supplementation (Experimental): Participants receive curcumin 390 mg combined with piperine 20 mg daily for 28 consecutive days following primary percutaneous coronary intervention (PPCI) for ST-elevation myocardial infarction (STEMI). A loading dose of 2 capsules (each containing 390 mg curcumin + 20 mg piperine) is administered orally prior to PPCI, followed by maintenance of 1 capsule daily until day 28.
  Interventions: Dietary Supplement: Curcumin plus Piperine

INTERVENTIONS:
Dietary Supplement: Curcumin plus Piperine — A loading dose of 2 capsules (each containing 390 mg curcumin + 20 mg piperine) is administered orally prior to PPCI, followed by maintenance of 1 capsule daily until day 28. Oral administration of standardized curcumin extract (390 mg) combined with piperine (20 mg), given twice daily for 28 days in addition to standard-of-care therapy for STEMI patients undergoing primary percutaneous coronary intervention (PPCI). The curcumin-piperine formulation is used to enhance bioavailability and anti-inflammatory effects, aiming to improve post-MI recovery and reduce oxidative stress.
  Other Names: Curcuma Xanthorrhiza with Piper Nigrum; Turmeric Extract with Piperine
  Arms: Curcumin-Piperine Supplementation
Other: Placebo capsules — A loading dose of 2 capsules (each containing saccarum lactic) is administered orally prior to PPCI, followed by maintenance of 1 capsule daily until day 28. Oral administration of standardized placebo capsule, given twice daily for 28 days in addition to standard-of-care therapy for STEMI patients undergoing primary percutaneous coronary intervention (PPCI).
  Arms: Placebo

SUMMARY:
This study aims to evaluate whether supplementation with a combination of curcumin and piperine can help reduce inflammation and oxidative stress in patients who have experienced a heart attack called ST-Elevation Myocardial Infarction (STEMI) and are undergoing a procedure known as primary percutaneous coronary intervention (PPCI).

Curcumin, a natural compound from turmeric, is known for its antioxidant and anti-inflammatory effects, but it is not easily absorbed by the body. Piperine, a compound from black pepper, can improve curcumin absorption. By combining the two, we hope to maximize their potential benefits.

The study will measure markers of inflammation (high-sensitivity C-reactive protein, hsCRP) and oxidative stress (malondialdehyde, MDA) at three time points: before treatment, shortly after the PPCI procedure, and after 28 days of supplementation.

The main question is whether curcumin-piperine supplementation can provide additional protection against inflammation and oxidative stress compared to a placebo, potentially supporting recovery and reducing the risk of future heart problems.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical trial investigates the effects of combined curcumin and piperine supplementation on systemic inflammation and oxidative stress in patients with ST-Elevation Myocardial Infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI). Curcumin, the principal curcuminoid derived from Curcuma xanthorrhiza or Curcuma longa, has demonstrated anti-inflammatory and antioxidant properties in preclinical and clinical studies. However, its oral bioavailability is limited due to poor absorption and rapid metabolism. Piperine, an alkaloid from Piper nigrum, enhances curcumin's bioavailability through inhibition of hepatic and intestinal glucuronidation.

Participants are randomized to receive either curcumin-piperine supplementation (390 mg curcumin + 20 mg piperine daily) or matched placebo for 28 consecutive days post-PPCI. Biomarkers of inflammation (high-sensitivity C-reactive protein, hsCRP) and oxidative stress (malondialdehyde, MDA) are assessed at three predefined time points: baseline (pre-intervention), 48-72 hours after PPCI, and at day 28 post-supplementation.

The primary objective is to determine whether curcumin-piperine supplementation significantly attenuates the rise in hsCRP and MDA levels compared to placebo. Secondary objectives include evaluating the temporal pattern of biomarker changes and assessing the tolerability and safety profile of the supplementation in the acute and subacute phases post-STEMI. The findings may provide evidence for adjunctive nutraceutical therapy to improve post-MI recovery by targeting inflammatory and oxidative stress pathways.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years.
* Confirmed diagnosis of ST-Elevation Myocardial Infarction (STEMI). Symptom onset within 12 hours, or within 12 to 72 hours in cases with an indication for primary percutaneous coronary intervention (PPCI).
* Receiving standard-of-care medical therapy according to current guidelines, including:

Dual antiplatelet therapy. Angiotensin-Converting Enzyme Inhibitors (ACE-i) or Angiotensin Receptor Blockers (ARBs).

Statins. Beta-blockers.

Exclusion Criteria:

* Regular prior use of curcumin supplementation.
* Hemodynamic instability or severe dyspnoea with clinical signs of congestion (elevated jugular venous pressure, pulmonary rales affecting >1/3 of lung fields, hepatomegaly, ascites, or peripheral oedema).
* History of prior myocardial infarction, previous percutaneous coronary intervention, or coronary artery bypass graft surgery.
* Known hypersensitivity to curcumin or piperine.
* Active malignancy.
* Chronic infections (e.g., hepatitis, tuberculosis, or HIV).
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m² or rapidly declining renal function.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Serum High-Sensitivity C-Reactive Protein (hsCRP) at Day 28 | Baseline (pre-intervention), within 48-72 hours post-PPCI and after 28 days of intervention
  Mean change (Δ) in serum hsCRP from baseline to Day 28, expressed in mg/L. Lower values indicate less systemic inflammation. The prespecified metric is group-wise mean change and between-group difference in mean change.
Change from Baseline in Malondialdehyde (MDA) at Day 28 | Baseline (pre-intervention), within 48-72 hours post-PPCI and after 28 days of intervention
  Mean change (Δ) in serum MDA concentration from baseline to Day 28, expressed in nmol/mL. Lower values indicate less lipid peroxidation/oxidative stress. The prespecified metric is group-wise mean change and between-group difference in mean change.

SECONDARY OUTCOMES:
Liver Function | Baseline and after 28 days of intervention
  To assess changes in liver enzyme activity (ALT and AST) as a marker of hepatic safety and potential hepatoprotective effect of curcumin-piperine supplementation. Unit of Measure: U/L.
Change in Serum Creatinine Levels | Baseline and after day 28 of intervention
  Serum creatinine will be measured to evaluate kidney function at baseline and after 28 days of supplementation. Unit of Measure: mg/dL.
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline and after day 28 of intervention
  eGFR will be calculated using the CKD-EPI formula to assess kidney function at baseline and after 28 days of supplementation. Unit of Measure: mL/min/1.73 m².

CONTACTS AND LOCATIONS:
Overall Officials: Fahri Husaini Alkaf, M.D., Principal Investigator — Universitas Diponegoro
Locations (1):
- Universitas Diponegoro, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The IPD will not be made publicly available due to ethical restrictions and confidentiality agreements with participants, as approved by the institutional review board.

REFERENCES:
- [Background] Lao CD, Ruffin MT 4th, Normolle D, Heath DD, Murray SI, Bailey JM, Boggs ME, Crowell J, Rock CL, Brenner DE. Dose escalation of a curcuminoid formulation. BMC Complement Altern Med. 2006 Mar 17;6:10. doi: 10.1186/1472-6882-6-10. PMID 16545122
- [Background] Soni KB, Kuttan R. Effect of oral curcumin administration on serum peroxides and cholesterol levels in human volunteers. Indian J Physiol Pharmacol. 1992 Oct;36(4):273-5. PMID 1291482
- [Background] Shacham Y, Leshem-Rubinow E, Gal-Oz A, Ben-Assa E, Steinvil A, Keren G, Roth A, Arbel Y. Relation of in-hospital serum creatinine change patterns and outcomes among ST-segment elevation myocardial infarction patients undergoing primary percutaneous coronary intervention. Clin Cardiol. 2015 May;38(5):274-9. doi: 10.1002/clc.22384. Epub 2015 Feb 1. PMID 25639761
- [Background] Trujillo J, Chirino YI, Molina-Jijon E, Anderica-Romero AC, Tapia E, Pedraza-Chaverri J. Renoprotective effect of the antioxidant curcumin: Recent findings. Redox Biol. 2013 Sep 17;1(1):448-56. doi: 10.1016/j.redox.2013.09.003. PMID 24191240
- [Background] Shoskes D, Lapierre C, Cruz-Correa M, Muruve N, Rosario R, Fromkin B, Braun M, Copley J. Beneficial effects of the bioflavonoids curcumin and quercetin on early function in cadaveric renal transplantation: a randomized placebo controlled trial. Transplantation. 2005 Dec 15;80(11):1556-9. doi: 10.1097/01.tp.0000183290.64309.21. PMID 16371925
- [Background] Albert MA, Staggers J, Chew P, Ridker PM; PRINCE Investigators. The pravastatin inflammation CRP evaluation (PRINCE): rationale and design. Am Heart J. 2001 Jun;141(6):893-8. doi: 10.1067/mhj.2001.115297. PMID 11376301
- [Background] Wongcharoen W, Jai-Aue S, Phrommintikul A, Nawarawong W, Woragidpoonpol S, Tepsuwan T, Sukonthasarn A, Apaijai N, Chattipakorn N. Effects of curcuminoids on frequency of acute myocardial infarction after coronary artery bypass grafting. Am J Cardiol. 2012 Jul 1;110(1):40-4. doi: 10.1016/j.amjcard.2012.02.043. Epub 2012 Apr 3. PMID 22481014
- [Background] Boshagh K, Khorvash F, Sahebkar A, Majeed M, Bahreini N, Askari G, Bagherniya M. The effects of curcumin-piperine supplementation on inflammatory, oxidative stress and metabolic indices in patients with ischemic stroke in the rehabilitation phase: a randomized controlled trial. Nutr J. 2023 Dec 11;22(1):69. doi: 10.1186/s12937-023-00905-1. PMID 38082237
- [Background] Panahi Y, Hosseini MS, Khalili N, Naimi E, Majeed M, Sahebkar A. Antioxidant and anti-inflammatory effects of curcuminoid-piperine combination in subjects with metabolic syndrome: A randomized controlled trial and an updated meta-analysis. Clin Nutr. 2015 Dec;34(6):1101-8. doi: 10.1016/j.clnu.2014.12.019. Epub 2015 Jan 7. PMID 25618800
- [Background] El-Saadony MT, Yang T, Korma SA, Sitohy M, Abd El-Mageed TA, Selim S, Al Jaouni SK, Salem HM, Mahmmod Y, Soliman SM, Mo'men SAA, Mosa WFA, El-Wafai NA, Abou-Aly HE, Sitohy B, Abd El-Hack ME, El-Tarabily KA, Saad AM. Impacts of turmeric and its principal bioactive curcumin on human health: Pharmaceutical, medicinal, and food applications: A comprehensive review. Front Nutr. 2023 Jan 10;9:1040259. doi: 10.3389/fnut.2022.1040259. eCollection 2022. PMID 36712505
- [Background] Singgih Wahono C, Diah Setyorini C, Kalim H, Nurdiana N, Handono K. Effect of Curcuma xanthorrhiza Supplementation on Systemic Lupus Erythematosus Patients with Hypovitamin D Which Were Given Vitamin D3 towards Disease Activity (SLEDAI), IL-6, and TGF-beta1 Serum. Int J Rheumatol. 2017;2017:7687053. doi: 10.1155/2017/7687053. Epub 2017 Dec 28. PMID 29445400
- [Background] Cai X, Fang Z, Dou J, Yu A, Zhai G. Bioavailability of quercetin: problems and promises. Curr Med Chem. 2013;20(20):2572-82. doi: 10.2174/09298673113209990120. PMID 23514412
- [Background] Pizzino G, Irrera N, Cucinotta M, Pallio G, Mannino F, Arcoraci V, Squadrito F, Altavilla D, Bitto A. Oxidative Stress: Harms and Benefits for Human Health. Oxid Med Cell Longev. 2017;2017:8416763. doi: 10.1155/2017/8416763. Epub 2017 Jul 27. PMID 28819546
- [Background] Moller P, Wallin H, Knudsen LE. Oxidative stress associated with exercise, psychological stress and life-style factors. Chem Biol Interact. 1996 Sep 27;102(1):17-36. doi: 10.1016/0009-2797(96)03729-5. PMID 8827060
- [Background] Shoba G, Joy D, Joseph T, Majeed M, Rajendran R, Srinivas PS. Influence of piperine on the pharmacokinetics of curcumin in animals and human volunteers. Planta Med. 1998 May;64(4):353-6. doi: 10.1055/s-2006-957450. PMID 9619120
- [Background] Liu W, Zhai Y, Heng X, Che FY, Chen W, Sun D, Zhai G. Oral bioavailability of curcumin: problems and advancements. J Drug Target. 2016 Sep;24(8):694-702. doi: 10.3109/1061186X.2016.1157883. Epub 2016 Mar 17. PMID 26942997
- [Background] Aggarwal BB, Sundaram C, Malani N, Ichikawa H. Curcumin: the Indian solid gold. Adv Exp Med Biol. 2007;595:1-75. doi: 10.1007/978-0-387-46401-5_1. PMID 17569205
- [Background] Abe Y, Hashimoto S, Horie T. Curcumin inhibition of inflammatory cytokine production by human peripheral blood monocytes and alveolar macrophages. Pharmacol Res. 1999 Jan;39(1):41-7. doi: 10.1006/phrs.1998.0404. PMID 10051376
- [Background] Mehta A, Blumenthal RS, Gluckman TJ, Feldman DI, Kohli P. High-sensitivity C-reactive Protein in Atherosclerotic Cardiovascular Disease: To Measure or Not to Measure? US Cardiol. 2025 Mar 21;19:e06. doi: 10.15420/usc.2024.25. eCollection 2025. PMID 40171210
- [Background] Wrobel-Nowicka K, Wojciechowska C, Jachec W, Zalewska M, Romuk E. The Role of Oxidative Stress and Inflammatory Parameters in Heart Failure. Medicina (Kaunas). 2024 May 2;60(5):760. doi: 10.3390/medicina60050760. PMID 38792942
- [Background] Neuhof C, Neuhof H. Calpain system and its involvement in myocardial ischemia and reperfusion injury. World J Cardiol. 2014 Jul 26;6(7):638-52. doi: 10.4330/wjc.v6.i7.638. PMID 25068024
- [Background] Mensah GA, Fuster V, Roth GA. A Heart-Healthy and Stroke-Free World: Using Data to Inform Global Action. J Am Coll Cardiol. 2023 Dec 19;82(25):2343-2349. doi: 10.1016/j.jacc.2023.11.003. No abstract available. PMID 38092508
- [Background] Martins-Marques T, Coutinho G, Kiss A. Editorial of the Special Issue: Cellular Mechanisms of Cardiovascular Disease. Biomedicines. 2023 Sep 8;11(9):2494. doi: 10.3390/biomedicines11092494. PMID 37760934
- [Background] GBD 2017 Causes of Death Collaborators. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1736-1788. doi: 10.1016/S0140-6736(18)32203-7. Epub 2018 Nov 8. PMID 30496103